CLINICAL TRIAL: NCT03414190
Title: Impact of a Mobile Phone Text Messages Intervention on the Secondary Prevention of Cardiovascular Events After Acute Coronary Syndrome
Brief Title: Impact of Text Messages to Promote Secondary Prevention After Acute Coronary Syndrome
Acronym: IMPACS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Antonio Luiz Pinho Ribeiro, Principal Investigator, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CEP1.883.227
Record Dates: First submitted 2018-01-14; First posted 2018-01-29 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Cardiovascular Disease
Keywords: Acute Coronary Syndrome; Text Messaging; Risk Factors
MeSH Terms: conditions — Cardiovascular Diseases; Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Automated semi-personalized mobile phone text message-based intervention for secondary prevention plus usual care.
  Interventions: Behavioral: Mobile phone text message
- No Intervention (No Intervention): Usual Care

INTERVENTIONS:
Behavioral: Mobile phone text message — The treatment group will receive the usual discharge treatment, instructions and information for acute coronary syndrome patients as well as the text-messaging intervention. The program will include a variety of topics such as standard follow-up care reminders as well as general self-management and healthy living habits texts. There will be four streams: one for patients who are non-smokers and are free of diabetes; one for current/recent smokers; one for diabetic patients; and one for smoker and diabetic patients. Texts will be sent out 4 times per week for 180 days. All participants in the same stream will receive the same texts in the same order. The usual care group will receive standard discharge treatment, instructions, and information for patients with acute coronary syndrome. They will also receive simple and short text messages related to the importance of trial participation.
  Arms: Experimental

SUMMARY:
The study is a two-arm, parallel, randomized clinical trial. The purpose of the study is to evaluate the effectiveness of automated mobile phone text message-based intervention for secondary prevention after acute coronary syndrome hospitalization. Text messages will include information about lifestyle modifications, medication adherence and cardiovascular risk factor control. The participants will be randomized into intervention and control groups in a 1:1 ratio. The intervention group will receive 4 pre-designed and semi-personalized text messages per week in addition to usual care for 6 months, while the control group will receive usual care.

DETAILED DESCRIPTION:
Purpose of the trial: The purpose of the study is to evaluate the effectiveness of automated mobile phone text message-based intervention for secondary prevention after acute coronary syndrome hospitalization.

Trial design: Two-parallel arm, single-blind, block randomization.

Primary endpoint: The proportion achieving guideline levels of modifiable risk factors (LDL-C <70mg/dL, blood pressure <140/90 mm Hg, exercising regularly [≥5 d/wk × 30minutes of moderate exercise per session], nonsmoker status, and BMI <25). The investigators prespecified in the statistical analysis plan the efficacy variable of proportion achieving combined risk factor control (achieving risk factor targets in 4 or more of the 5 modifiable risk factors listed above) as a measure of a multiple risk factor effect.

Secondary endpoints: The plasma LDL-C level at 6 months, Level of physical activity, Blood Pressure, Medication adherence measured via Morisky scale, Proportion of non-smokers, Body mass index (BMI), Rates death and hospitalization up to 6 months.

Duration of follow-up: 6 months

Trial treatment:

Intervention: The treatment group will receive the usual discharge treatment, instructions and information for acute coronary syndrome patients as well as the text-messaging intervention. The program will include a variety of topics such as standard follow-up care reminders as well as general self-management and healthy living habits texts. There will be four streams: one for patients who are non-smokers and are free of diabetes; one for current/recent smokers; one for diabetic patients; and one for smoker and diabetic patients. Texts will be sent out 4 times per week for 180 days. All participants in the same stream will receive the same texts in the same order.

Control: The usual care group will receive standard discharge treatment, instructions, and information for patients with acute coronary syndrome. The participants will also receive SMS thanking for their participation in the trial, reminders of trial appointment and informing if they have changed contact details. The frequency of this SMS will be monthly.

Expected sample size, enrollment and expected number of centers:

Sample size = 160 Recruitment start date: November, 2017 Recruitment end date: May, 2019 Follow-up end date: November, 2019 Number of centers: 1

Statistical considerations:

* Intention to treat analysis
* The trial has >90% power (2 sided alpha = 0.05) to detect 15% difference in achieving risk factor targets in 4 or more of the 5 modifiable risk factors listed.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients who have been hospitalized at the UFMG's University Hospital with primary or secondary diagnosis of Acute Coronary Syndrome and are discharged for outpatient follow-up;
* Age ≥ 18 years, of both sexes;
* Patients who are able to receive text messages by their own mobile phone.

Exclusion Criteria:

* Refusal or inability to sign the Informed Consent.
* Complete illiteracy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2017-11-29 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Escore of combined risk factor control | 6 months
  The proportion achieving guideline levels of modifiable risk factors (LDL-C <77mg/dL, blood pressure <140/90 mm Hg, exercising regularly [≥5 d/wk × 30minutes of moderate exercise per session], nonsmoker status, and BMI <25). We prespecified in the statistical analysis plan the efficacy variable of proportion achieving combined risk factor control (achieving risk factor targets in 4 or more of the 5 modifiable risk factors listed above) as a measure of a multiple risk factor effect

SECONDARY OUTCOMES:
Plasma LDL-C level | 6 months
  Fasting blood sample
Level of physical activity (measured via | 6 months
  Measured by research blinded to treatment allocation - The level of physical activity will be mensured by the International Physical Activity Questionnaire Short Form (IPAQ-SF) and it will be validated in one-fifth of the participants by using accelerometers
Blood Pressure | 6 months
  Measured by research blinded to treatment allocation - 3 resting, sitting digital recordings, mean of last 2 readings
Proportion of non-smokers | 6 months
  Measured by research blinded to treatment allocation - Self-reported smoking / quitting attempts will be confirmed with a Carbon Monoxide Meter Breath Test
Body mass index (BMI) | 6 months
  Measured by research blinded to treatment allocation
Medication adherence (measured via "Medida de adesão aos tratamentos" - MAT) | 6 months
  Measured by research blinded to treatment allocation It is an instrument composed of seven items that evaluate the behavior of the individual in relation to daily use of medicines. The answers are obtained by means of a six-point ordinal scale that varies from always (1) to never (6). The values obtained with the answers to the seven items are summed and divided by the number of items (values vary from 1 to 6). Subsequently, values 5 and 6 are computed as one (adherent) and the others are computed as zero (non-adherent).
Death from any cause | 6 months
  Medical records and database
Rehospitalization | 6 months
  Self-report, medical records and database
Cardiovascular death | 6 months
  Medical records and database

CONTACTS AND LOCATIONS:
Locations (1):
- Luiz Guilherme Passaglia, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No